CLINICAL TRIAL: NCT05103189
Title: 4D Flow Cardiac MRI Velocity Mapping in Patients With Pulmonary Hypertension: Estimation of Pulmonary Arterial Pressure and Comparison With Right Heart Catheterization and Doppler Echocardiography
Brief Title: 4D-flow Cardiac MRI to Assess Pulmonary Arterial Pressure in Pulmonary Hypertension
Acronym: HTPFLUW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2020_843_0062
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Hypertension; Magnetic Resonance Imaging; Pulmonary Arterial Pressure; Right Heart Catheterization; Echocardiography
Keywords: Pulmonary Hypertension; 4D-flow magnetic resonance imaging; mean pulmonary arterial pressure; right heart catheterization; echocardiography
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 4D-flow sequence — all patients will be referred for a complete cardiac MRI exam with the addition of a 4D Flow sequence (does not require supplementary injection of a contrast agent and does not extend the duration of the examination) followed promptly (within the same hour) by a Doppler-echocardiography.

SUMMARY:
Due to radiation exposure and low but real risk of morbidity and mortality associated with right heart catheterization, non-invasive procedures to estimate mPAP are desired for the diagnosis of PH or to monitor treatment effectiveness. Echocardiography is used as a screening tool to estimate systolic pulmonary arterial pressure (sPAP), but due various limitations, this technique is not considered to be sufficiently accurate for the diagnosis of PH. The aim of 4D flow MRI is to evaluate the complete time-varying tridirectional velocity field in a volume of interest. It enables flow and velocity measurements in a vascular region of interest and visualization of vector plots of blood flow velocity fields. Previous studies have shown on the one hand, correlations between mPAP and hemodynamic parameters obtained by phase contrast MRI and, on the other hand, appearance of a vortical blood flow in the pulmonary artery in PH. More studies are required to confirm 4D MRI as a valuable tool for mPAP estimation in PH.

Following screening echocardiography, all patients will undergo right heart catheterization for PH assessment. Then, all patients will be referred for a complete cardiac MRI exam with the addition of a 4D Flow sequence (does not require supplementary injection of a contrast agent and does not extend the duration of the examination) followed promptly (within the same hour) by a Doppler-echocardiography. The data from each examination will be blindly interpreted from the results of the other one. No follow-up will be required for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Patient referred for cardiac MRI who previously underwent right heart catheterization for pulmonary hypertension assessment,
* Affiliation to a social security program,
* Ability of the subject to understand and express opposition

Exclusion Criteria:

* Age <18 years old,
* Major obesity (> 140 kg) not allowing the patient to enter the tunnel of the machine whose diameter is less than 70 cm,
* Person under guardianship or curators,
* Pregnant woman,
* Allergy to gadolinium chelates,
* Claustrophobia,
* Any contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between the values of mPAP (mmHg) and right heart catheterization rate. | 30 minutes
  mPAP is obtained by 4D flow MRI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No